CLINICAL TRIAL: NCT04876963
Title: HOLT-ED: Holter-monitoring in End-stage Renal Disease - Does Burden of Arrhythmia Assessed With Systematic Holter Electrocardiogram Monitoring Affect Cardiovascular Outcomes? - A Prospective Cohort Study
Brief Title: HOLT-ED: Holter-monitoring in End-stage Renal Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicholas Carlson, MD PhD, Rigshospitalet, Denmark
Other Study IDs: HOLT-ED protocol 1.10
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Kidney Failure, Chronic; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Holter-monitor — 7-day holtermonitoring of each patient

SUMMARY:
The main objective of this prospective cohort study is to assess arrhythmia burden and glycemic variability in a multicenter cohort of patients with end-stage renal disease using a sufficient observation period in order to identify arrhythmia burden and type and characterize associations with patient characteristics and dialysis treatment, glycemic variability and subsequent risk of adverse outcomes.

DETAILED DESCRIPTION:
Background: The risk of dying of a cardiovascular disease is 10-20 times increased in patients dependent on dialysis treatment compared to the general population. 1/3 of these deaths is caused by arrhythmia and 'sudden cardiac death'.

Purpose: Investigate the prevalence and type of arrhythmia in patients dependent on dialysis treatment, including the association with patient- and dialysis related factors and cardiovascular outcomes.

Methods: 7-days Holter-monitoring with Cortrium C3+ holter-monitor in 540 patients dependent on dialysis treatment in the Capital Region of Denmark. Continous blood glucose monitoring in a subgroup. 1-year follow-up via national registers.

Endpoints:

* Prevalence of atrial fibrillation
* Prevalence of other arrhythmia (tachycardia, bradycardia, AV-block)
* Follow-up outcomes: sudden cardiac death, cardiovascular disease and cardiovascular death

ELIGIBILITY:
Inclusion Criteria:

* Dialysis-treated end-stage renal disease
* Age ≥ 18 years
* Competence to understand the study rationale necessary for written informed consent

Exclusion Criteria:

* Pre-existing pacemaker implantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with dialysis-treated end-stage renal disease over the age of 18 and without pacemaker implantation.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-05 (Estimated); Study Completion 2024-09-05 (Estimated)

PRIMARY OUTCOMES:
Sudden cardiac death / lethal arrhythmia | 1-year follow up
  Risk of sudden cardiac death or lethal arrhythmia within one year
Cardiovascular death | 1-year follow up
  Risk of cardiovascular death within one year
All-cause mortality | 1-year follow up
  Risk of all-cause mortality within one year
Myocardial infarction or death attributable to myocardial infarction | 1-year follow up
  Risk of Myocardial infarction or death attributable to myocardial infarction within one year

OTHER OUTCOMES:
Clinical hypoglycemia | Baseline
  Clinical hypoglycemia in connection with holtermonitoring at baseline
De novo cardiac arrhythmia (atrial fibrillation or flutter, advanced second-degree or third degree | Baseline
  De novo cardiac arrhythmia (atrial fibrillation or flutter, advanced second-degree or third degree at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Carlson, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Dept. of Nephrology, Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - North Zealand Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
Tabulated study data and protocols will be made available (within limitations of Danish legislation related to GDPR)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: within 1 year of study completion
Access Criteria: Data access will be available upon approval via Statistics Denmark